CLINICAL TRIAL: NCT03526094
Title: Flavanol Absorption, Metabolism and Excretion From Fruit-based Drinks and Other Food Matrixes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 429275-D
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: flavanol; ADME; polyphenols; Cocoa; Banana; epicatechin

STUDY DESIGN:
Intervention Model Description: Cross-over dietary intervention study in healthy young adult males
Who Masked: Investigator
Masking Description: Investigator processing samples and performing statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Flavanols-capsules (Active Comparator): Capsules containing 541 mg cocoa flavanols (75 mg epicatechin) and 315 g of milk (1% fat)
  Interventions: Other: Flavanols-capsules
- Flavanol-banana blend (Experimental): Fruit blend prepared by mixing 177 g ripe, frozen bananas, 240 g almond milk and a chocolate flavored powder containing 638 mg cocoa flavanols (88 mg epicatechin)
  Interventions: Other: Flavanol-banana blend
- Flavanol-high protein drink (Experimental): Drink prepared by mixing 225 mL of a chocolate flavored high protein dairy drink with a CF powder containing 565 mg cocoa flavanols (78 mg epicatechin)
  Interventions: Other: Flavanol-high protein drink
- Flavanol-berry blend (Experimental): Fruit blend prepared by mixing 120 g almond milk, 70 g water, 95 g yogurt, 50 g each strawberries, blueberries, blackberries, raspberries, 105 g crushed ice and a fruit-flavored powder containing 484 mg cocoa flavanols (68 mg epicatechin)
  Interventions: Other: Flavanol-berry blend
- Flavanol-sports drink (Experimental): Drink prepared by mixing 488 g of a sports drink with a CF powder containing 565 mg cocoa flavanols (78 mg epicatechin)
  Interventions: Other: Flavanol-sports drink
- Flavanol-peanut butter toast (Experimental): Prepared by mixing 32 g peanut butter with a chocolate flavored powder containing 653 mg cocoa flavanols (85 mg epicatechin) and spread on 1 slice toasted bread (50 g) and 50 g sliced strawberries
  Interventions: Other: Flavanol-peanut butter toast
- Flavanol-oats (Experimental): Prepared by mixing 40 g quick oats with 237 g boiling water and combined with a chocolate flavored powder containing 653 mg cocoa flavanols (85 mg epicatechin)
  Interventions: Other: Flavanol-oats
- Flavanol-yogurt (Experimental): Prepared by 227 g yogurt (0% fat) mixed with a fruit-flavored powder containing 484 mg cocoa flavanols (68 mg epicatechin)
  Interventions: Other: Flavanol-yogurt
- II- Flavanol drink (Active Comparator): Drink prepared by mixing 240 g almond milk with a chocolate flavored powder containing 638 mg cocoa flavanols (88 mg epicatechin)
  Interventions: Other: II- Flavanol drink
- II- Flavanol drink + banana blend (Experimental): Drink 1 (Flavanol drink): prepared by mixing 120 g almond milk with 638 mg cocoa flavanols (88 mg epicatechin) Drink 2 (Fruit blend): prepared by mixing 120 g almond milk blended with 177 g ripe, frozen bananas
  Interventions: Other: II- Flavanol drink + banana blend

INTERVENTIONS:
Other: Flavanols-capsules — Capsules containing 456 mg cocoa flavanols and 315 g of milk (1% fat)
  Arms: Flavanols-capsules
Other: Flavanol-banana blend — Fruit blend prepared by mixing 177 g ripe, frozen bananas, 240 g almond milk and a chocolate flavored powder containing 626 mg cocoa flavanols
  Arms: Flavanol-banana blend
Other: Flavanol-high protein drink — Drink prepared by mixing 225 mL of a chocolate flavored high protein dairy drink with a CF powder containing 533 mg cocoa flavanols
  Arms: Flavanol-high protein drink
Other: Flavanol-berry blend — Flavanol-berry blend prepared by mixing 120 g almond milk, 70 g water, 95 g yogurt, 50 g each strawberries, blueberries, blackberries, raspberries, 105 g crushed ice and a fruit-flavored powder containing 561 mg cocoa flavanols
  Arms: Flavanol-berry blend
Other: Flavanol-sports drink — Drink prepared by mixing 488 g of a sports drink with a CF powder containing 533 mg cocoa flavanols
  Arms: Flavanol-sports drink
Other: Flavanol-peanut butter toast — Prepared by mixing 32 g peanut butter with a chocolate flavored powder containing 602 mg cocoa flavanols and spread on 1 slice toasted bread (50 g) and 50 g sliced strawberries
  Arms: Flavanol-peanut butter toast
Other: Flavanol-oats — Prepared by mixing 40 g quick oats with 237 g boiling water and combined with a chocolate flavored powder containing 602 mg cocoa flavanols
  Arms: Flavanol-oats
Other: Flavanol-yogurt — Prepared by 227 g yogurt (0% fat) mixed with a fruit-flavored powder containing 561 mg cocoa flavanols
  Arms: Flavanol-yogurt
Other: II- Flavanol drink — Drink prepared by mixing 240 g almond milk with a chocolate flavored powder containing 626 mg cocoa flavanols
  Arms: II- Flavanol drink
Other: II- Flavanol drink + banana blend — Drink 1 (Flavanol drink): prepared by mixing 120 g almond milk with 626 mg cocoa flavanols Drink 2 (Fruit blend): prepared by mixing 120 g almond milk blended with 177 g ripe, frozen bananas
  Arms: II- Flavanol drink + banana blend

SUMMARY:
Dietary intervention study in healthy adult males to evaluate concentration of flavanol metabolites in plasma and urine after single acute intakes of flavanols from different fruit-based drinks.

DETAILED DESCRIPTION:
Flavonoids, including the sub groups of Flavanols (F) are plant-derived compounds commonly present in the human diet. Examples of F-containing foods and beverages are apples, chocolate, tea, wine, berries, pomegranate and nuts. The consumption of F-containing foods and beverages has been associated with improvements in cardiovascular health. In this context, there exists a great interest in describing the absorption, metabolism and excretion of F in humans, as it is thought that F-derived metabolites present in circulation are the mediators of F-beneficial effects in humans. Recently, the investigators described a series of F-derived metabolites in circulation that are present after the consumption of a single acute intake amount of F in humans as well as F-metabolites derived from the metabolic activity of the gut microbiome. A key question, however, is if the metabolites we observed after a single acute feeding are the same as those that occur in individuals who consume F-rich diets on a regular basis. Studies investigating the metabolism of numerous other xenobiotics have shown that the profile of metabolites can greatly vary over time, as well as with the amount of the xenobiotic ingested. In this context, the investigators submit it is important to assess whether or not there are food matrix-dependent effects on the levels and profile of F-derived metabolites in humans. The investigators suggest the information that will be obtained from the outlined work will be particularly timely given ongoing discussion concerning the possible generation of dietary recommendations for F-rich foods and increasing interest in the putative health effects of F intake in humans.

This study consisted of two parts. One part investigated flavanols absorption and metabolism from different fruit-based drinks and other food matrixes. The second part investigated flavanol absorption and metabolism after the intake of a flavanol drink alone and simultaneously consumed with a banana-based drink.

Following the beginning of the trial, an advanced method to analyze cocoa flavanols was accredited by AOAC International as a First Action Official Method of Analysis https://doi.org/10.1093/jaoacint/qsaa132). This updated method relies on a reference material (RM8403) recently standardized and made commercially available by the U.S. National Institute of Standards and Technology. While the actual cocoa flavanol content of our intervention remained unchanged throughout the trial, the application of this new analytical method led to expected changes in how the total cocoa flavanol content is now reported. Applying AOAC 2020.05/RM8403 to our intervention, the total cocoa flavanol content of select arms in our trials have been updated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* No prescription medications
* BMI 18.5 - 29.9 kg/m2
* Weight ≥ 110 pounds
* previously consumed cocoa, peanut, parsley, celery and chamomile products with no adverse reactions

Exclusion Criteria:

* Adults unable to consent
* Prisoners
* Non-English speaking*
* BMI ≥ 30 kg/m2
* Performing vigorous physical activity (i.e. more than 6 MET; metabolic equivalence of task as defined by CDC and ACSM guidelines (http://www.cdc.gov/physicalactivity/everyone/glossary/index.html#vig-intensity; and http://www.cdc.gov/nccdphp/dnpa/physical/pdf/PA_Intensity_table_2_1.pdf ) for more than 3 days a week.
* Dietary allergies including those to nuts, cocoa and chocolate products, parsley, celery and chamomile.
* Active avoidance of coffee and caffeinated soft drinks
* Under current medical supervision
* A history of cardiovascular disease, stroke, renal, hepatic, or thyroid disease
* History of clinically significant depression, anxiety or other psychiatric condition
* History of Raynaud's disease
* History of difficult blood draws
* Indications of substance or alcohol abuse within the last 3 years
* Current use of herbal, plant or botanical supplements (multi-vitamin/mineral supplements are allowed)
* Blood Pressure > 140/90 mm Hg
* GI tract disorders, previous GI surgery (except appendectomy)
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Diarrhea within the last 3 months, or antibiotic intake within the last 3 months
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individuals following diets with significant deviations from the average diet
* Metabolic panel and cholesterol results or complete blood counts that are outside of the normal reference range and are considered clinically relevant by the study physician
* Cold, flu, or upper respiratory condition at screening
* Currently participating in a clinical or dietary intervention study

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Flavanol metabolites in plasma | Before to 6 h post test material intake
  Plasma concentration of flavanol metabolites

SECONDARY OUTCOMES:
Flavanol metabolites in urine | 12 h before to 24 h post test material intake
  Amount of flavanols metabolites excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis; Javier I Ottaviani, PhD, Study Director — Mars, Inc.
Locations (2):
- United States (2):
  - Ragle Human Nutrition Research Center, Department of Nutrition at UC Davis, Davis, California
  - UC Davis, Davis, California

IPD SHARING:
Plan to Share IPD: Yes
Only researchers listed in the protocol and approved by the IRB will have access to IPD.

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838
- [Background] Ottaviani JI, Momma TY, Kuhnle GK, Keen CL, Schroeter H. Structurally related (-)-epicatechin metabolites in humans: assessment using de novo chemically synthesized authentic standards. Free Radic Biol Med. 2012 Apr 15;52(8):1403-12. doi: 10.1016/j.freeradbiomed.2011.12.010. Epub 2011 Dec 23. PMID 22240152
- [Background] Koster H, Halsema I, Scholtens E, Knippers M, Mulder GJ. Dose-dependent shifts in the sulfation and glucuronidation of phenolic compounds in the rat in vivo and in isolated hepatocytes. The role of saturation of phenolsulfotransferase. Biochem Pharmacol. 1981 Sep 15;30(18):2569-75. doi: 10.1016/0006-2952(81)90584-0. No abstract available. PMID 6946775
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Heiss C, Kleinbongard P, Dejam A, Perre S, Schroeter H, Sies H, Kelm M. Acute consumption of flavanol-rich cocoa and the reversal of endothelial dysfunction in smokers. J Am Coll Cardiol. 2005 Oct 4;46(7):1276-83. doi: 10.1016/j.jacc.2005.06.055. PMID 16198843